CLINICAL TRIAL: NCT05263479
Title: A Phase I, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of HS-20089 in Patients With Advanced Solid Tumors
Brief Title: A Study of HS-20089 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hansoh Biomedical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Hansoh BioMedical R&D Company (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20089-101
Record Dates: First submitted 2021-10-29; First posted 2022-03-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor
Keywords: HS-20089; ADC; B7-H4; Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20089 (Phase Ia：Dose escalation ) (Experimental): HS-20089 for IV infusion of various dose strengths administered in 21 day dosing cycles.
  Interventions: Drug: HS-20089 (Phase Ia：Dose escalation )
- HS-20089 (Phase Ib: Dose expansion) (Experimental): The recommended dose from the dose-escalation stage and other potential doses will be further explored.
  Interventions: Drug: HS-20089 (Phase Ib: Dose expansion)

INTERVENTIONS:
Drug: HS-20089 (Phase Ia：Dose escalation ) — Participants will receive HS-20089 in 21 day dosing cycles. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Arms: HS-20089 (Phase Ia：Dose escalation )
Drug: HS-20089 (Phase Ib: Dose expansion) — IV administration of HS-20089 Q3W; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
  Arms: HS-20089 (Phase Ib: Dose expansion)

SUMMARY:
HS-20089 is a novel DAR-6 antibody-drug conjugate （ADC） targeting B7-H4. In preclinical studies, it inhibited tumor cell growth expressing B7-H4 in vitro and in vivo. The first-in-human trial is conducted to assess the maximum tolerated dose (MTD) and dose limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of HS-20089 in Patients With Advanced Solid Tumors.

DETAILED DESCRIPTION:
This is a Phase 1a/1b open-label, multicenter study with dose escalation and dose expansion cohorts to evaluate the safety, tolerability, PK and preliminary efficacy of HS-20089 in patients with advanced solid tumors.

The Dose Escalation will include an initial accelerated titration design followed by a Bayesian optimal interval (BOIN) design. Enrollment into Dose Expansion will begin after identification of the MTD and/or MAD in Phase 1a. In Phase 1b, preliminary efficacy will be evaluated in planned expansion cohorts that include patients with specific tumor types that are B7-H4+ advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years
2. Advanced solid tumor patients confirmed by histology or cytology for who that standard treatment is invalid, unavailable or intolerable
3. Patients have at least one target lesion according to RECEST 1.1. The requirements for target lesions are: measurable lesions without local treatment such as irradiation, or with definite progress after local treatment, with the longest diameter ≥ 10 mm in the baseline period (in case of lymph nodes, the shortest axis ≥ 15 mm is required)
4. ECOG performance status was 0-1 and did not deteriorate in the previous 2 weeks
5. Estimated life expectancy greater than (>) 12 weeks
6. Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have evidence of non-childbearing potential
7. Sign Informed Consent Form

Exclusion Criteria:

1. Treatment with any of the following:

   1. Previous or current treatment with drugs targeting B7-H4
   2. Any cytotoxic chemotherapy, investigational agents or anticancer drugs within 28 days of the first dose of study drug
   3. Radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study drug, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks of the first dose.
   4. Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) within 4 weeks of the first dose of study drug.
   5. Known and untreated, or active central nervous system metastases.
2. Existing abnormal CTCAE≥grade 2 resulted from previous treatment
3. History of other malignancy
4. Inadequate bone marrow reserve or organ function
5. Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV), unless the hepatitis is considered to be cured, Known history of HIV
6. History of hypersensitivity to any active or inactive ingredient of HS-20089.
7. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
8. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of HS-20089 | 3 weeks after initiation of treatment
  To determine the MTD for further evaluation of IV administration of HS-20089 in subjects with advanced solid tumors.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | Baseline through study completion(90 days after last dose)
  The CTCAE criteria will be used to assess adverse events on this trial.
Observed maximum plasma concentration (Cmax) after single dose of HS-20089 | From pre-dose to 120 hours after single dose on Day 1
  Cmax will be obtained after single dose of HS-20089 on Day 1.
Observed maximum plasma concentration (Cmax ss) after multiple dose of HS-20089 | From pre-dose to 24 hours after the dose on Day 1 of the 21-Day cycle of therapy
  Cmax ss will be obtained on Day 1 of dosing in the 21-Day cycle of therapy.
Apparent terminal half-life (t1/2) after single dose of HS-20089 | From pre-dose to 120 hours after single dose on Day 1
  Apparent terminal half-life is the time measured for the concentration to decrease by one half.
Area under plasma concentration versus time curve from zero to the 24-hour sampling time (AUC0-24) after single dose of HS-20089 | From pre-dose to 24 hours after single dose on Day 1
  Area under the plasma concentration versus time curve from time zero to the 24-hour sampling time at which the concentration was at or above the lower limit of quantification (LLQ).
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) after single dose of HS-20089 | From pre-dose to 120 hours after single dose on Day 1
  Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ).
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) after single dose of HS-20089 | From pre-dose to 120 hours after single dose on Day 1
  AUC0-∞ was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the LLQ and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
To further evaluation of the anti-tumor activity of HS-20089 by assessment of objective response rate (ORR) | From the date of first occurrence of complete response (CR) or partial response (PR) on 2 consecutive occasions (≥4 weeks), until the date of disease progression or withdrawal from study，up to 2 years
  Anti-tumor efficacy will be assessed by best radiographic response based on Response Evaluation Criteria in Solid Tumors at baseline (Day -28 to -1). For patients that continue on repeating 21-Day cycles after the primary evaluation period, progression will be assessed after each 6 weeks of therapy. ORR is defined as the percentage of patients with a complete response (CR) or partial response (PR) that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.
Anti-drug Antibodies (ADA) of HS-20089 | Baseline through study completion(90 days after last dose)
  Number of participants who test positive for ADA to HS-20089 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No